CLINICAL TRIAL: NCT03716037
Title: Improving Physical and Psychosocial Well-being of African American Older Adults Living in Rural Areas Through a Community-Based Exercise Program
Brief Title: Improving Physical and Psychosocial Well-being of African American Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Principal Investigator, Mercy N. Mumba, Assistant Professor, University of Alabama, Tuscaloosa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-010-ME
Record Dates: First submitted 2018-10-11; First posted 2018-10-23 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Physical Activity; Psychosocial Stressors
Keywords: physical activity; exercise; depression; anxiety; stress
MeSH Terms: conditions — Motor Activity; Depression; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): Physical Activity for Life (PAL) is an 8-week exercise program, meeting three times per week for one hour sessions.
  Interventions: Other: Physical Activity for Life (PAL)
- Contact Control (No Intervention): those in the attentional contact control group will receive a phone call from research personnel three times per week asking them about their physical exercise routines.

INTERVENTIONS:
Other: Physical Activity for Life (PAL) — The eight-week exercise program (The PAL Study) will incorporate balance, strength, endurance, and flexibility training. The duration of each exercise session, which will be offered three times a week, will be one hour. The supervised exercise session will include 30 minutes of moderate-intensity aerobic exercise, 15 minutes of resistance training, and 15 minutes of stretching and balance training
  Arms: Physical Activity

SUMMARY:
The proposed research effort will:

The purpose of this study is as follows:

1. Test the feasibility and acceptability of an eight-week community-based exercise program among AA older adults living in rural areas.
2. Determine whether participation in physical exercise through a community-based exercise program in comparison with an attentional control group: a) improves physical well-being b) improves psychosocial well-being

DETAILED DESCRIPTION:
Among the aging population, African Americans (AA) experience depression and other chronic diseases such as diabetes, hypertension, and cardiovascular disease at a higher rate compared to non-minorities; moreover, those living in rural areas are less likely to seek treatment due to various factors including lack of accessibility, affordability, and acceptability of health care services. Fortunately, non-pharmacologic and cost-effective interventions such as physical activity can yield physical, psychosocial, and cognitive benefits for older adults. The purpose of the proposed research effort is to test the feasibility of, and effect of a community-based physical exercise program among community-dwelling older adults living in rural areas on the physical and psychosocial well-being. The research effort will be a randomized controlled trial. Fifty African American older adults will be recruited from community centers. A total of 50 participants will be recruited. These adults will be randomly assigned to either the intervention or control group, with each group containing 25 participants. The intervention will occur over a period of eight week. The exercise program will be offered three times a week, with each session lasting one hour. Study measures will be collected prior to the start of the exercise program, after the fourth session, after the last session, and at one-month follow-up. The primary outcome measures for the feasibility study will include enrollment rate, randomization rate, retention rate, and data completion rate. Additionally, the investigators will examine whether there is improvement I both physical and psychosocial measures. All statistical analyses will be conducted using Statistical Package for the Social Sciences (SPSS) version 22.

ELIGIBILITY:
Inclusion Criteria:

1. At least 65 years of age
2. Identifying as AA
3. community dwelling and living in a rural community.
4. Sedentary life style (engaging in less than two hours of structured physical exercises whether independently or in a group setting every week)
5. Identify as having altered psychosocial health by scoring at least a 10 on the Patient Health Questionnaire (PHQ-9), which is indicative of moderate depressive symptoms (Kroenke, Spitzer, & Williams, 2001).

Exclusion Criteria:

1. cognitive impairment as defined by the St. Louis University Mental Status Exam

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the community based exercise program as measured by enrollment rate | 12 months
  enrollment rate which is the number of participants who sign the informed consent form divided by the number who are approached should be ≥ 60%

SECONDARY OUTCOMES:
physical activity as measured by Fitbit trackers | 12 months
  Fitbit will track the daily steps
psychosocial Well-being as measured by the Patient Reported Outcomes Measurement Information Systems (PROMIS) Global Health Measure-10 | 12 months
  Primary psychosocial variables of interest, that is depression and anxiety will be measured using the PROMIS Global Health Measure-10, a 10-item questionnaire that examines physical, mental, and social health. The questions focus on the previous seven days. This tool is scored on a 5-point Likert scale. Internal consistency of the subscales ranges from Cronbach's alpha = 0.8-0.92. Scores range from 10-50. Higher values indicate higher functioning for all scales- physical, mental or social scales.
Satisfaction Outcome as measured by the Client satisfaction Questionnaire | 12 months
  Satisfaction with the intervention program will be assessed with the 8-item Client Satisfaction Questionnaire (CSQ-8; Attkisson, 2012), with established reliability, internal consistency, and validity across racial/ethnic groups. Summary scores range from 8-32 with higher scores indicating greater satisfaction. Study-specific satisfaction items will be assessed also using a 4-pt Likert scale . Higher scores mean increased participant satisfaction.
Physical Function as measured by the senior fitness test | 12 months
  all seven components of the senior fitness test will be examined. This is a validated tool for physical function in older adults.
physical activity as measured by Fitbit trackers | 12 months
  Fitbit will track number of minutes active every day.
Feasibility of the community based exercise program as measured by randomization rate | 12 months
  randomization rate which is the number of participants randomized divided by the number of participants consented and screened which should be ≥ 60%
Feasibility of the community based exercise program as measured by retention rate | 12 months
  retention rate which is the number of participants completing T2 divided by the number who were randomized should be ≥ 80%.

CONTACTS AND LOCATIONS:
Overall Officials: Mercy N Mumba, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Uniontown Recreation Center, Uniontown, Alabama, United States

IPD SHARING:
Plan to Share IPD: No